CLINICAL TRIAL: NCT01940835
Title: Role of Intestinal Inflammation in the Pathogenesis of Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); University of Chicago (Other); Harvard University (Other)
Responsible Party: Principal Investigator, Joseph A. Murray, M.D., Professor of Medicine, Mayo Clinic
Other Study IDs: 12-003972
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Gastroscopy; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, DNA, RNA extraction, brush biopsies from duodenal mucosa, biopsies of small intestine, stool samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Type 1 Diabetes: Subjects will have an upper endoscopy with small bowel biopsies and brushings. Blood will be collected for serum, DNA, and peripheral blood mononuclear cells (PBMC). Stool samples will be collected at baseline for future microbiome and virome studies.
  Interventions: Procedure: Upper endoscopy with small bowel biopsies and brushings.; Other: Blood draw; Other: Stool sample
- Healthy Control Group: Subjects will have an upper endoscopy with small bowel biopsies and brushings. Blood will be collected for serum, DNA, and peripheral blood mononuclear cells (PBMC). Stool samples will be collected at baseline for future microbiome and virome studies.
  Interventions: Procedure: Upper endoscopy with small bowel biopsies and brushings.; Other: Blood draw; Other: Stool sample

INTERVENTIONS:
Procedure: Upper endoscopy with small bowel biopsies and brushings.
Other: Blood draw — Blood will be collected for serum, DNA, and peripheral blood mononuclear cells (PBMC).
Other: Stool sample — Stool samples will be collected at baseline for future microbiome and virome studies.

SUMMARY:
This purpose of this study is to determine if activation of a person's immune system in the small intestine could be a contributing cause of Type 1 Diabetes.

DETAILED DESCRIPTION:
There is a large body of literature hinting at a role of the gut in Type One Diabetes (T1D) pathogenesis. However, to the best of our knowledge there is no definitive evidence to date conclusively demonstrating a link. The only way to test this hypothesis is to have access to the intestinal tissue of T1D patients at very early stages when beta-islet cell destruction is still ongoing. Furthermore, to prepare for large prospective studies it is critical to determine whether there is a peripheral blood signature for intestinal inflammation. Finally, because enteroviral infections have been implicated in T1D pathogenesis, this study provides a unique opportunity to determine whether there is a dysregulated response to innate stimuli associated with viral infections and whether evidence of transcriptional signatures indicative of viral infections in the gut is correlated with disease. Finally, we will take advantage of this pilot study to collect samples that can be used for microbiome, virome and metabolic studies.

ELIGIBILITY:
For the Diabetes Cohort:

Inclusion Criteria:

* Initial diagnosis for Type 1 Diabetes Mellitus (DM) must be within the past 6 months.
* Clinical criteria used to diagnose T1D include at least some of the following : Diabetic ketoacidosis, Polyuria, Polydipsia, weight loss, need for insulin from diagnosis, BMI less than 30, C-peptide < 200 pmol/L or 0.6 ng/ml, Presence of Type 1 Diabetes Associated Antibodies

Exclusion Criteria:

* Subjects on antibiotics, proton pump inhibitors, aspirin, non-steroidal anti-inflammatory drugs, alcohol intake within 48 hours, a bowel preparation with 4 weeks of the studies, and smokers
* Subjects will be asked not to take any probiotics in the week before testing.
* Any known intestinal inflammation such as Gastroesophageal Reflux Disease (GERD), eosinophilic esophagitis, and inflammatory bowel disease.
* Prior gastrointestinal surgery (other than appendectomy)
* Ongoing use of antiplatelet agents or anticoagulants.
* Diabetic patients should not have a prior history of or family history of Celiac Disease (CD).
* Subjects unable to provide informed consent
* The presence of any medical or psychological condition that could interfere with the safe performance of the upper endoscopy.
* Females cannot be pregnant

For the Healthy Control Cohort:

Inclusion Criteria:

- Healthy subjects

Exclusion Criteria:

* Controls should not have a family history of DM or CD
* Subjects on antibiotics, proton pump inhibitors, aspirin, non-steroidal anti-inflammatory drugs, alcohol intake within 48 hours, a bowel preparation with 4 weeks of the studies, and smokers
* Subjects will be asked not to take any probiotics in the week before testing.
* Any known intestinal inflammation such as Gastroesophageal Reflux Disease (GERD), eosinophilic esophagitis, and inflammatory bowel disease.
* Prior gastrointestinal surgery (other than appendectomy)
* Ongoing use of antiplatelet agents or anticoagulants.
* Subjects unable to provide informed consent
* The presence of any medical or psychological condition that could interfere with the safe performance of the upper endoscopy.
* Females cannot be pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Type 1 Diabetes, diagnosed within 6 months
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
Mean Interleukin 15 (IL-15) Expression | baseline, 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Murray, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials